CLINICAL TRIAL: NCT00998062
Title: Dyslipaemia, Atherosclerosis Risk and Increased hsCRP and Inflammatory and Oxidative Status in the Spanish Population
Brief Title: Dyslipaemia, Atherosclerosis Risk and Increased hsCRP and Inflammatory and Oxidative Status in the Spanish Population. Database Analysis of Previous Studies Performed in Spain
Acronym: DARIOS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CES-DUM-2009/1
Record Dates: First submitted 2009-10-19; First posted 2009-10-20 (Estimated); Last update posted 2011-10-20 (Estimated); Status verified 2011-10

CONDITIONS: Dyslipaemia; Atherosclerosis Risk; Increased hsCRP; Inflammatory and Oxidative Status in the Spanish Population
Keywords: Dyslipaemia; atherosclerosis risk; increased hsCRP; inflammatory and oxidative status in the Spanish population

STUDY DESIGN:
Time Perspective: Retrospective
Biospecimen Retention: None Retained — No samples will be obtained, but biomarkers will be analysed from frozen serum samples retained by the pervious studies performed.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Data from epidemiological studies performed after the year 2000 with patients between 35 and 74 years old

SUMMARY:
The present project is aimed at determining the prevalence of LDL-C <130 mg/dl with hsCRP ≥2mg/l, and of HDL-C < 40 mg/dl in Spain together with the estimation of cardiovascular risk, to analyze the contribution of measuring hsCRP for primary prevention purposes. In a subgroup of that population a number of inflammatory and oxidative status biomarkers would be also measured to better understand the meaning of elevated hsCRP.The study aim to analyze data already collected in studies (11 studies will participate) carried out in Spain, in 10 Spanish regions, after the year 2000.

ELIGIBILITY:
Inclusion Criteria:

* Have an Informed consent form signed when the patient accepted to participate in the study already performed.
* Spanish population between
* Data from Epidemiological studies performed after the year 2000

Exclusion Criteria:

* Spanish population outside the age range
* Data from Epidemiological studies performed before the year 2000

Ages: 35 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data from epidemiological studies performed after the year 2000 with patients between 35 and 74 years old
Sampling Method: Probability Sample
Enrollment: 30181 (Estimated)
Dates: Start 2009-11; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Lipid fractions: high-density lipoprotein, low-density lipoprotein, and total cholesterol, and triglycerides, and dislipidemia treatments | retrospectively

SECONDARY OUTCOMES:
High sensitivity C reactive protein & CHR risk by Framingham adapted functions | retrospectively
Lipid profile among the Spanish regions, as in the primary outcome variable | retrospectively
Biomarkers: Interleukines 6 and 10, oxidized LDL, VCAM, ICAM, TNF alpha, neopterin, fibrinogen, lp(a), MMP 9 Apo A, Apo B, adiponectin, leptin, resistin, and yet other | prospectively

CONTACTS AND LOCATIONS:
Locations (11):
- Spain (11):
  - Research Site, Andalucia, Andalusia
  - Research Site, Canarias, Canary Islands
  - Research Site, Castilla Y Leon, Castille and León
  - Research Site, Talavero, Castille-La Mancha
  - Research Site, Girona, Catalonia
  - Research Site, Hospitalet, Catalonia
  - Research Site, Badajoz, Extremadura
  - Research Site, Madrid, Madrid
  - Research Site, Mallorca, Mallorca
  - Research Site, Murcia, Murcia
  - Research Site, Navarra, Navarre